CLINICAL TRIAL: NCT03844685
Title: RED CLOVER EXTRACT (PROMENSIL) AND LIFESTYLE CHANGES TO CONTRAST MENOPAUSAL SYMPTOMS IN PREMENOPAUSAL WOMEN WITH HORMONE-SENSITIVE BREAST CANCER RECEIVING ADJUVANT ANTI-ESTROGEN THERAPY
Brief Title: Red Clover and Lifestyle Changes to Contrast Menopausal Symptoms in Premenopausal Breast Cancer Patients Given Tamoxifen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INT 101/11
Record Dates: First submitted 2018-12-20; First posted 2019-02-18 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Promensil

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient and personnel involved in trial masked to treatment vs. placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): 1 tablet /day of MCE-11 (Promensil) taken orally for 24 months
  Interventions: Drug: Promensil
- Placebo group (Placebo Comparator): Placebo tablet (without active principle) given once a day for 24 months
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Promensil — 1 tablet (80 mg) /day of MCE-11 (Promensil) taken orally for 24 months
  Arms: Treatment group
Drug: Placebo Oral Tablet — Placebo tablet (80 mg) (without active principle) given once a day for 24 months
  Arms: Placebo group

SUMMARY:
A prospective double-blind randomized trial of red clover extract (Promensil) vs placebo in surgically-treated premenopausal women with estrogen receptor-positive breast cancer taking tamoxifen

DETAILED DESCRIPTION:
Premenopausal women with ER-positive breast cancer treated by surgery and receiving postoperative tamoxifen with or without LHRH analogues, who may have received pre or postoperative chemotherapy, or immunotherapy (for HER2-positive disease), are recruited to a double-blind randomized clinical trial, to receive either a dry extract of red clover (Promensil) as one tablet/day orally containing 80 mg isoflavones (treatment group), or one oral tablet/day without active principle (placebo group) for 24 months. All patients receive a diet-lifestyle intervention involving meetings with a dietician (physician) scheduled once a month for the first 6 months, and every 3 months thereafter. The dietician encourages patients to adhere to a macronutrient-balanced, low glycaemic load Mediterranean-type diet with personalized recommendations to increase intakes of unrefined cereals, pulses, vegetables, unrefined vegetable fats (e.g. olive oil, nuts, oil-containing seeds), and fish, and reduce intake of high-glycaemic-index foods and saturated animal fats. Patients are also encouraged to undertake regular physical activity. Outcomes are Menopausal Rating Score (MRS), body mass index (BMI), waist and hip girth, insulin resistance, and levels of cholesterol, triglycerides, and sex hormones.

The safety of the red clover preparation is assessed by pelvic ultrasound and mammograms for endometrial thickness and breast density, and by evaluation of the effects of the serum from treated and placebo patients on ER-positive BC cell lines.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed operable ER-positive breast cancer
* Can be ductal carcinoma in situ (DCIS)
* Absence of locoregional relapse or distant metastasis
* Normal ovarian function
* Menopause Rating Score > or equal to 8
* Signed informed consent to participate

Exclusion Criteria:

* Menopause Rating Score <8
* Menopausal at diagnosis or at surgery
* Previous malignancies other than in situ cervical carcinoma or non-melanoma skin cancer
* Breast cancer recurrence
* Metastatic breast cancer
* Non-epithelial breast cancer at histological examination
* In situ lobular breast cancer
* Participation in other randomized clinical trials that could interfere with current study
* Living distant from center and unable to attend for check-ups and meetings.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 88 (Actual)
Dates: Start 2012-07-05 (Actual); Primary Completion 2014-03-25 (Actual); Study Completion 2016-02-23 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) | 24 months
  Full name of questionnaire is "Menopause Rating Scale" ; The total score of the MRS ranges between 0 (asymptomatic) and 44 (highest degree of complaints). the ranges are: 0-4 no/little symptoms, 5-8 mild, 9-15 moderate and 16/16+ severe.
  The sub-scale are: Psychological score, (Question N° 4-7), Somatic score (Question N° 1-3; 11), Urogenital score (Question N° 8-10). The subscales are combined in a total MRS score.
weight gain (kg) | 24 months
insulin resistance | 24 months
  fasting blood glucose x fasting blood insulin (HOMA-IR)

SECONDARY OUTCOMES:
endometrial thickness | 24 months
  assessed by annual pelvic ultrasound (mm)
breast density | 24 months
  assessed by annual mammography (BI-RADS)
growth of breast cancer cell lines highly expressing estrogen receptors | 24 months
  OD Units
transcript expression of estrogen-regulated genes in breast cancer cell lines highly expressing estrogen receptors | 24 months
  transcript levels

CONTACTS AND LOCATIONS:
Locations (1):
- Cristina Ferraris, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dornstauder E, Jisa E, Unterrieder I, Krenn L, Kubelka W, Jungbauer A. Estrogenic activity of two standardized red clover extracts (Menoflavon) intended for large scale use in hormone replacement therapy. J Steroid Biochem Mol Biol. 2001 Jul;78(1):67-75. doi: 10.1016/s0960-0760(01)00075-9. PMID 11530286
- [Result] Piersen CE, Booth NL, Sun Y, Liang W, Burdette JE, van Breemen RB, Geller SE, Gu C, Banuvar S, Shulman LP, Bolton JL, Farnsworth NR. Chemical and biological characterization and clinical evaluation of botanical dietary supplements: a phase I red clover extract as a model. Curr Med Chem. 2004 Jun;11(11):1361-74. doi: 10.2174/0929867043365134. PMID 15180571
- [Result] Imhof M, Molzer S, Imhof M. Effects of soy isoflavones on 17beta-estradiol-induced proliferation of MCF-7 breast cancer cells. Toxicol In Vitro. 2008 Sep;22(6):1452-60. doi: 10.1016/j.tiv.2008.04.018. Epub 2008 May 4. PMID 18554862
- [Result] Howes J, Waring M, Huang L, Howes LG. Long-term pharmacokinetics of an extract of isoflavones from red clover (Trifolium pratense). J Altern Complement Med. 2002 Apr;8(2):135-42. doi: 10.1089/107555302317371424. PMID 12006121
- [Result] Kawakita S, Marotta F, Naito Y, Gumaste U, Jain S, Tsuchiya J, Minelli E. Effect of an isoflavones-containing red clover preparation and alkaline supplementation on bone metabolism in ovariectomized rats. Clin Interv Aging. 2009;4:91-100. doi: 10.2147/cia.s4164. Epub 2009 May 14. PMID 19503771
- [Result] Atkinson C, Compston JE, Day NE, Dowsett M, Bingham SA. The effects of phytoestrogen isoflavones on bone density in women: a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2004 Feb;79(2):326-33. doi: 10.1093/ajcn/79.2.326. PMID 14749241
- [Result] Lipovac M, Chedraui P, Gruenhut C, Gocan A, Stammler M, Imhof M. Improvement of postmenopausal depressive and anxiety symptoms after treatment with isoflavones derived from red clover extracts. Maturitas. 2010 Mar;65(3):258-61. doi: 10.1016/j.maturitas.2009.10.014. Epub 2009 Nov 30. PMID 19948385
- [Result] Imhof M, Gocan A, Reithmayr F, Lipovac M, Schimitzek C, Chedraui P, Huber J. Effects of a red clover extract (MF11RCE) on endometrium and sex hormones in postmenopausal women. Maturitas. 2006 Aug 20;55(1):76-81. doi: 10.1016/j.maturitas.2006.01.006. Epub 2006 Mar 2. PMID 16513301
- [Result] Hidalgo LA, Chedraui PA, Morocho N, Ross S, San Miguel G. The effect of red clover isoflavones on menopausal symptoms, lipids and vaginal cytology in menopausal women: a randomized, double-blind, placebo-controlled study. Gynecol Endocrinol. 2005 Nov;21(5):257-64. doi: 10.1080/09513590500361192. PMID 16373244
- [Result] Terzic MM, Dotlic J, Maricic S, Mihailovic T, Tosic-Race B. Influence of red clover-derived isoflavones on serum lipid profile in postmenopausal women. J Obstet Gynaecol Res. 2009 Dec;35(6):1091-5. doi: 10.1111/j.1447-0756.2009.001059.x. PMID 20144173
- [Result] Chedraui P, San Miguel G, Hidalgo L, Morocho N, Ross S. Effect of Trifolium pratense-derived isoflavones on the lipid profile of postmenopausal women with increased body mass index. Gynecol Endocrinol. 2008 Nov;24(11):620-4. doi: 10.1080/09513590802288283. PMID 19031218
- [Result] Mueller M, Jungbauer A. Red clover extract: a putative source for simultaneous treatment of menopausal disorders and the metabolic syndrome. Menopause. 2008 Nov-Dec;15(6):1120-31. doi: 10.1097/gme.0b013e31817062ce. PMID 18724264
- [Result] Simoncini T, Fornari L, Mannella P, Caruso A, Garibaldi S, Baldacci C, Genazzani AR. Activation of nitric oxide synthesis in human endothelial cells by red clover extracts. Menopause. 2005 Jan-Feb;12(1):69-77. doi: 10.1097/00042192-200512010-00013. PMID 15668603
- [Result] Teede HJ, McGrath BP, DeSilva L, Cehun M, Fassoulakis A, Nestel PJ. Isoflavones reduce arterial stiffness: a placebo-controlled study in men and postmenopausal women. Arterioscler Thromb Vasc Biol. 2003 Jun 1;23(6):1066-71. doi: 10.1161/01.ATV.0000072967.97296.4A. Epub 2003 Apr 24. PMID 12714433
- [Result] Guha N, Kwan ML, Quesenberry CP Jr, Weltzien EK, Castillo AL, Caan BJ. Soy isoflavones and risk of cancer recurrence in a cohort of breast cancer survivors: the Life After Cancer Epidemiology study. Breast Cancer Res Treat. 2009 Nov;118(2):395-405. doi: 10.1007/s10549-009-0321-5. Epub 2009 Feb 17. PMID 19221874
- [Result] Chlebowski RT, Schwartz AG, Wakelee H, Anderson GL, Stefanick ML, Manson JE, Rodabough RJ, Chien JW, Wactawski-Wende J, Gass M, Kotchen JM, Johnson KC, O'Sullivan MJ, Ockene JK, Chen C, Hubbell FA; Women's Health Initiative Investigators. Oestrogen plus progestin and lung cancer in postmenopausal women (Women's Health Initiative trial): a post-hoc analysis of a randomised controlled trial. Lancet. 2009 Oct 10;374(9697):1243-51. doi: 10.1016/S0140-6736(09)61526-9. Epub 2009 Sep 18. PMID 19767090
- [Result] Cross HS, Kallay E, Lechner D, Gerdenitsch W, Adlercreutz H, Armbrecht HJ. Phytoestrogens and vitamin D metabolism: a new concept for the prevention and therapy of colorectal, prostate, and mammary carcinomas. J Nutr. 2004 May;134(5):1207S-1212S. doi: 10.1093/jn/134.5.1207S. PMID 15113973
- [Result] Horn-Ross PL, John EM, Canchola AJ, Stewart SL, Lee MM. Phytoestrogen intake and endometrial cancer risk. J Natl Cancer Inst. 2003 Aug 6;95(15):1158-64. doi: 10.1093/jnci/djg015. PMID 12902445
- [Result] Horn-Ross PL, Hoggatt KJ, Lee MM. Phytoestrogens and thyroid cancer risk: the San Francisco Bay Area thyroid cancer study. Cancer Epidemiol Biomarkers Prev. 2002 Jan;11(1):43-9. PMID 11815400